CLINICAL TRIAL: NCT07348744
Title: The Effect of a Health Belief Model-Based Education Program on Breast Self-Examination Practice Behavior, Breast Cancer Fear, and Awareness Levels in Women: A Randomized Controlled Trial
Acronym: KAU-BSE-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Cansu Karadağ, Principal Investigator, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KAU-BSE-RCT
Record Dates: First submitted 2025-12-29; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Breast Self-Examination; Breast Cancer
Keywords: Breast Self-Examination; Breast Cancer; Health Belief Model
MeSH Terms: conditions — Breast Self-Examination; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to an intervention group receiving a Health Belief Model-based education program or to a control group receiving usual care.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to group allocation. Due to the nature of the educational intervention, participants and intervention providers are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Belief Model-Based Education Group (Experimental): Participants receive a structured education program based on the Health Belief Model focusing on breast self-examination.
  Interventions: Behavioral: Health Belief Model-Based Education Program
- Control Group (No Intervention): Participants receive usual care without any additional educational intervention.

INTERVENTIONS:
Behavioral: Health Belief Model-Based Education Program — A structured education program based on the Health Belief Model designed to improve breast self-examination behavior and increase breast cancer awareness.
  Arms: Health Belief Model-Based Education Group

SUMMARY:
The study titled "The Effect of a Health Belief Model-Based Training Program on Women's Self-Breast Examination Behavior, Breast Cancer Fear and Awareness Levels: A Randomized Controlled Study" aimed to increase breast cancer awareness and the application of breast self-examination techniques among women by providing the necessary training through a training program based on the Health Belief Model.

DETAILED DESCRIPTION:
This randomized controlled study aims to evaluate the effectiveness of a Health Belief Model-based education program on women's breast self-examination practices, breast cancer fear, and awareness levels. Participants will be randomly assigned to either an intervention group receiving a structured education program based on the Health Belief Model or a control group receiving usual care.

Data will be collected using a Personal Information Form, the Champion Health Belief Model Scale, the Comprehensive Breast Cancer Knowledge Test, the Breast Cancer Awareness Scale, and the Champion Breast Cancer Fear Scale at baseline and three months after the intervention. The findings of this study are expected to contribute to the development of effective educational strategies for improving breast cancer awareness and preventive health behaviors among women.

ELIGIBILITY:
Inclusion Criteria:

* Being affiliated with Family Health Center No. 1 in Ardahan Province,
* Being a woman between the ages of 20 and 69,
* Being literate,
* Not having been diagnosed with breast cancer,
* Not having a mental or communication disorder,
* Having a phone available for communication,
* Women who voluntarily agree to participate in the study.

Exclusion Criteria:

* Difficulty communicating,
* Wanting to drop out of the study,
* Not wanting to participate in the study.
* Women who did not fill out the data form despite reminders via message and phone call.

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Breast Self-Examination Behavior | Baseline and 3 months after the intervention
  Change in breast self-examination behavior measured as a single self-reported outcome indicating whether participants perform breast self-examination.

SECONDARY OUTCOMES:
Change in Breast Cancer Knowledge Level | Baseline and 3 months after the intervention
  Change in breast cancer knowledge assessed using the Comprehensive Breast Cancer Knowledge Test.
Change in Breast Cancer Awareness Level | Baseline and 3 months after the intervention
  Change in breast cancer awareness measured using the Breast Cancer Awareness Scale.
Change in Breast Cancer Fear Level | Baseline and 3 months after the intervention
  Change in fear related to breast cancer measured using the Champion Breast Cancer Fear Scale.

CONTACTS AND LOCATIONS:
Overall Officials: CANSU KARADAĞ, Principal Investigator — Kafkas University
Locations (1):
- Kafkas University, Kars, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No